CLINICAL TRIAL: NCT00443638
Title: Longitudinal Follow Up of Subjects Enrolled in Randomized Trials of Prenatal and Infancy Home Visitation
Brief Title: Longitudinal Follow Up of Subjects Enrolled in Randomized Trial of Prenatal and Infancy Home Visitation
Acronym: ElmiraY19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Smith-Richardson Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 98-0568
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Risk Reduction Behavior; Reproductive Behavior
MeSH Terms: conditions — Risk Reduction Behavior; Reproductive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): Control Group
- Home visitation through pregnancy (Experimental): Nurse home visitation through pregnancy
  Interventions: Behavioral: nurse home visitation
- Home visitation through age 2 (Experimental): Nurse home visitation through child age 2.
  Interventions: Behavioral: nurse home visitation

INTERVENTIONS:
Behavioral: nurse home visitation — Nurse home visitation
  Arms: Home visitation through age 2; Home visitation through pregnancy

SUMMARY:
The Elmira follow-up study is designed to assess the extent to which prenatal and infancy home visitation by nurses affects the life-course development of 19-year-old youth whose mothers received those services during pregnancy and the first two years of the child's life.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women prior to the 25th week of gestation
* no previous live births
* one of the following sociodemographic risk characteristics:

  * young age (< 19 years at registration);
  * unmarried
  * low socioeconomic status (Medicaid status or no private insurance)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 1998-05; Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
rates of pregnancy and out-of-wedlock child birth | At age 19
educational achievement, including graduation from high school and participation in various types of post-high school education | At age 19
participation in the work force, including enrollment in the armed services | At age 19
use of welfare | At age 19
use of substances (cigarettes, alcohol, and illegal drugs) | At age 19
involvement with the criminal justice system (arrests, convictions, incarcerations, etc.) | At age 19

CONTACTS AND LOCATIONS:
Overall Officials: David Olds, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- CIDS, Elmira, New York, United States

REFERENCES:
- [Background] Izzo CV, Eckenrode JJ, Smith EG, Henderson CR, Cole R, Kitzman H, Olds DL. Reducing the impact of uncontrollable stressful life events through a program of nurse home visitation for new parents. Prev Sci. 2005 Dec;6(4):269-74. doi: 10.1007/s11121-005-0010-5. PMID 16075193
- [Background] Eckenrode J, Zielinski D, Smith E, Marcynyszyn LA, Henderson CR Jr, Kitzman H, Cole R, Powers J, Olds DL. Child maltreatment and the early onset of problem behaviors: can a program of nurse home visitation break the link? Dev Psychopathol. 2001 Fall;13(4):873-90. PMID 11771912
- [Background] Eckenrode J, Ganzel B, Henderson CR Jr, Smith E, Olds DL, Powers J, Cole R, Kitzman H, Sidora K. Preventing child abuse and neglect with a program of nurse home visitation: the limiting effects of domestic violence. JAMA. 2000 Sep 20;284(11):1385-91. doi: 10.1001/jama.284.11.1385. PMID 10989400
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R. Intellectual impairment in children of women who smoke cigarettes during pregnancy. Pediatrics. 1994 Feb;93(2):221-7. PMID 8121734
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R. Prevention of intellectual impairment in children of women who smoke cigarettes during pregnancy. Pediatrics. 1994 Feb;93(2):228-33. PMID 7510063
- [Background] Olds DL, Henderson CR Jr, Kitzman H. Does prenatal and infancy nurse home visitation have enduring effects on qualities of parental caregiving and child health at 25 to 50 months of life? Pediatrics. 1994 Jan;93(1):89-98. PMID 8265329
- [Background] Olds DL, Henderson CR Jr, Phelps C, Kitzman H, Hanks C. Effect of prenatal and infancy nurse home visitation on government spending. Med Care. 1993 Feb;31(2):155-74. doi: 10.1097/00005650-199302000-00006. PMID 8433578
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R, Chamberlin R. Improving the life-course development of socially disadvantaged mothers: a randomized trial of nurse home visitation. Am J Public Health. 1988 Nov;78(11):1436-45. doi: 10.2105/ajph.78.11.1436. PMID 3052116
- [Background] Olds DL, Henderson CR Jr, Chamberlin R, Tatelbaum R. Preventing child abuse and neglect: a randomized trial of nurse home visitation. Pediatrics. 1986 Jul;78(1):65-78. PMID 2425334
- [Derived] Lane C, Hogg E, Karwatowska LA, French L, Ranieri VF, Jesnick LGD, Roberts C, Scott S, Senior R, Skinner GC, Kennedy EMM. Personalised interventions for subgroups of children with conduct problems. Cochrane Database Syst Rev. 2023 Apr 28;4(4):CD012746. doi: 10.1002/14651858.CD012746.pub2. PMID 37115724
- [Derived] Eckenrode J, Campa M, Luckey DW, Henderson CR Jr, Cole R, Kitzman H, Anson E, Sidora-Arcoleo K, Powers J, Olds D. Long-term effects of prenatal and infancy nurse home visitation on the life course of youths: 19-year follow-up of a randomized trial. Arch Pediatr Adolesc Med. 2010 Jan;164(1):9-15. doi: 10.1001/archpediatrics.2009.240. PMID 20048236